CLINICAL TRIAL: NCT04031547
Title: Functional MRI Study of Transcranial Electrical Stimulation in Major Depression
Brief Title: fMRI Study of tES in Major Depression
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Amber Leaver, Research Assistant Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STU00207022
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tES-fMRI (Active Comparator)
  Interventions: Device: Transcranial Electrical Stimulation (tES)
- Inactive/Sham tES-fMRI (Sham Comparator)
  Interventions: Device: Transcranial Electrical Stimulation (tES)

INTERVENTIONS:
Device: Transcranial Electrical Stimulation (tES) — In tES, a mild electrical current is passed between two or more electrodes placed on the scalp.
  Other Names: Transcranial Direct Current Stimulation (tDCS)

SUMMARY:
This is a functional MRI study that will examine the effects of noninvasive transcranial electrical stimulation (tES) on brain function in individuals with Major Depression.

DETAILED DESCRIPTION:
The purpose of this research study is to understand how a kind of brain stimulation, called transcranial electrical stimulation (tES), affects brain function in people with major depression.

tES delivers low electrical current to the head using electrodes applied to the skin, and is described as a "neuromodulation" or "neurostimulation" technique. This study uses a specific kind of tES called "transcranial direct current stimulation", or tDCS, where a constant (unchanging) electrical current is passed between two electrodes on the head.

Neuromodulation methods like tES have shown promise in changing brain function, as well as treating some brain disorders like major depression. Yet, how tES brain function remains unclear. To better understand how tES works, the investigators will use MRI (a type of brain scan) to measure brain function during tES in people with major depression.

ELIGIBILITY:
Inclusion Criteria:

* ages between 18 and 55
* diagnosis of Major Depressive Disorder made by a physician, psychiatrist, or psychologist at least one year prior
* mild-to-moderate symptoms of depression (Hamilton Depression Rating Scale 17-item, HDRS-17, score 8-23)
* stable standard or no pharmacological antidepressant regimen (SSRI, SNRI, MAOI, or trycyclic/TCA) with no change in treatment 6 weeks prior to study start

Exclusion Criteria:

* suicidal thoughts, ideation, or behavior within the past month (HDRS-17 item 3 score greater than 1)
* greater than moderate symptoms of depression within the past month (HDRS-17 score >23)
* change in antidepressant medication within 6 weeks of study start
* diagnosis of any medical condition potentially affecting brain function, including neuropsychiatric or mental disorders, other mood disorders (bipolar disorder, anxiety, PTSD), psychotic states or disorders, developmental disorders, neurological disorders, including mild cognitive impairment, significant head injury, significant history of alcohol/substance abuse or dependence
* MRI contraindications: metal or other implants that are not MR-safe, claustrophobia, pregnancy or suspected pregnancy
* tES contraindications: skin conditions or injuries on the scalp, hair extensions, wigs, braids, etc. that cannot be removed prior to the study, metal implants or pacemakers
* other major medical conditions (e.g., cancer, stroke)
* current medication use potentially affecting brain function, including decongestants, antihistamines, benzodiazepines or other anticonvulsants, anti-psychotics, or antidepressants
* prisoners will not participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in brain function measured with blood-oxygenation-level-dependent (BOLD) functional MRI | 5 minutes before, 5 minutes during, and 5 minutes after tES
  Blood-oxygenation-level-dependent functional MRI will be used to measure changes in the temporal coherence (functional connectivity) amongst brain regions before, during, and after tES.

CONTACTS AND LOCATIONS:
Overall Officials: Amber Leaver, PhD, Principal Investigator — Northwestern University
Locations (1):
- Center for Translational Imaging at Northwestern University, Chicago, Illinois, United States